CLINICAL TRIAL: NCT05634200
Title: Utility of Bronchoscopy in Patients With Haemoptysis and Negative Chest CT Scan: an Observational, Prospective, Multicentre Study (ULYSSES)
Brief Title: Utility of Bronchoscopy in Patients With Haemoptysis and Negative Chest CT Scan (ULYSSES)
Status: Recruiting | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Mondoni, Associate Professor of Respiratory Medicine, University of Milan
Other Study IDs: BrHaemoCTNeg
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hemoptysis
Keywords: Computed tomography; Bronchoscopy; Lung cancer; CT scan; Haemoptysis
MeSH Terms: conditions — Hemoptysis; Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, serum, bronchial/lung tissue, bronchial secretions, BAL fluid, lymph node aspirates
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haemoptysis and negative/non-diagnostic CT scan: Patients with haemoptysis and negative/non-diagnostic CT scan (i.e. with focal peripheral lung fibrosis, calcified parenchymal nodules with a maximum diameter <5 mm, linear subsegmental atelectasis, hilar-mediastinal lymph nodes with a short axis <1 cm, pleural thickening/pleural calcification and focal area of emphysema with a diameter <1 cm) for whom bronchoscopy is deemed necessary to obtain an aetiological diagnosis.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — During bronchoscopy endobronchial biopsy, transbronchial biopsy, transbronchial needle aspiration, bronchial washing, bronchoalveolar lavage, EBUS-TBNA and EUS-B-FNA may be performed

SUMMARY:
Conflicting evidence exist in the literature on the utility of bronchoscopy in patients with haemoptysis and negative/non-diagnostic chest CT scan.

The primary aim of this prospective, observational, multicenter study is to evaluate the utility of bronchoscopy in patients with haemoptysis and negative/non-diagnostic CT scans. Secondary aims are related to the utility of bronchoscopy to detect occult malignancies, the source of the bleeding and the clinical features of the cohort

DETAILED DESCRIPTION:
Haemoptysis, i.e., coughing up blood from the airways, is a common and alarming symptom in the context of respiratory diseases. Studies conducted in Europe and North America in the last ten years have identified lung cancer (13.9-30.3%), bronchiectasis (6-21%) and low respiratory tract infection (4.2-40%) as the most common causes of the symptom. No international guidelines exist suggesting the optimal diagnostic work-up in patients with haemoptysis, based on demographics characteristics, risk factors (such as smoking history) and clinical presentation. The full diagnostic pathway of the symptom includes patient anamnesis, blood tests, chest X-ray, chest computed tomography (CT) scan and bronchoscopy. The 2020 international guidelines of American College of Radiology recommends performing chest CT scan with intravenous (IV) contrast or a CT angiography after the first episode of haemoptysis of any severity. Many studies recommend CT scan before bronchoscopy, underlining the diagnostic complementarity of the tests and the role of tCT as a guide for endoscopic examination. There is conflicting evidence in the literature on the utility of bronchoscopy in patients with a negative CT scan or in cases of CT showing non-specific or non-diagnostic benign findings (e.g., calcified parenchymal nodule, linear subsegmental atelectasis, pleural thickening). Due to this conflicting evidence, we deem necessary to conduct a prospective, observational, multicentre study. The primary aim is to evaluate the proportion of patients with haemoptysis and negative/non-diagnostic CT scans in whom bronchoscopy allows an aetiological (i.e., endoscopic and/or microbiological and/or anatomopathological) diagnosis.

The secondary objectives are:

* to evaluate the proportion of patients in whom bronchoscopy may detect occult endobronchial neoplasms (not detected with chest CT scan)
* to evaluate the proportion of patients in whom bronchoscopy may identify the source of the bleeding
* to evaluate the proportion of patients with haemoptysis and negative chest CT scan in whom bronchoscopic findings may induce variation in the treatment of the patients
* to evaluate the proportion of patients with a negative bronchoscopy at baseline, in whom a subsequent endoscopic examination performed during the follow-up for recurrent haemoptysis may allow an aetiological (endoscopic and/or microbiological and/or anatomopathological) diagnosis
* to evaluate the proportion of patients with negative CT scan and bronchoscopy in whom lung cancer may be diagnosed during the follow-up
* to evaluate the main clinical characteristics (e.g., severity, duration of haemoptysis) of patients with haemoptysis with negative chest CT scan and bronchoscopy, the rate and severity of symptom recurrence and the mortality rate after one year of follow-up in this cohort.

The study will be performed in twelve Respiratory Units throughout Europe. The study will last two years, and it is estimated to enroll at least 150 adult patients of any nationality referred for haemoptysis of unknown origin with negative/non-diagnostic chest CT scan, for whom bronchoscopy is deemed necessary to obtain an aetiological diagnosis. Patients will undergo pulmonary examination and blood tests (complete blood count, PT, PTT, urea, blood creatinine and CRP) before bronchoscopy. A chest CT scan with IV contrast is considered necessary, except for patients with absolute contraindications (renal failure, allergy to iodinate IV contrast). Only patients with chest CT scan performed within 72 hours from the last episode of haemoptysis will be enrolled in the study. Bronchoscopy will be performed within two weeks of the chest CT scan. All the enrolled patients will be followed-up for 12 months with a telephone interview at one, three, six and twelve months after the enrolment. In case of haemoptysis relapse, a clinical evaluation could be performed. Each centre will decide upon the subsequent diagnostic work-up.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Haemoptysis of unknown origin
* Negative or non-diagnostic chest CT scan

Exclusion Criteria:

* Known bleeding lesions of the upper or lower respiratory airways
* Chest CT scan diagnostic for hemoptysis etiology
* Refusal to sign the informed consent
* Refusal of bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (i.e., ≥18 years) of any nationality (inpatients and outpatients) with haemoptysis of unknown aetiology and negative chest CT scan/with CT scan showing non-diagnostic findings (i.e. focal peripheral lung fibrosis, calcified parenchymal nodules with a maximum diameter <5 mm, linear subsegmental atelectasis, hilar-mediastinal lymph nodes with a short axis <1 cm, pleural thickening/pleural calcification and focal area of emphysema with a diameter <1 cm), in whom bronchoscopy is deemed necessary to obtain an aetiological diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of patients with haemoptysis and negative/non-diagnostic CT scans in whom bronchoscopy allows an aetiological (i.e., endoscopic and/or microbiological and/or anatomopathological) diagnosis | One year
  The primary aim of the study is to evaluate the proportion of patients with haemoptysis and negative/non-diagnostic CT scans in whom bronchoscopy allows an aetiological (i.e., endoscopic and/or microbiological and/or anatomopathological) diagnosis

SECONDARY OUTCOMES:
To evaluate the proportion of patients in whom bronchoscopy may detect occult endobronchial neoplasms (not detected with chest CT scan) | One year
  To evaluate the proportion of patients in whom bronchoscopy may detect occult endobronchial neoplasms (not detected with chest CT scan)
To evaluate the proportion of patients in whom bronchoscopy may identify the source of the bleeding | One year
  To evaluate the proportion of patients in whom bronchoscopy may identify the source of the bleeding
To evaluate the proportion of patients with haemoptysis and negative chest CT scan in whom bronchoscopic findings may induce variation in the treatment of the patients | One year
  To evaluate the proportion of patients with haemoptysis and negative chest CT scan in whom bronchoscopic findings may induce variation in the treatment of the patients
To evaluate the proportion of patients with a negative bronchoscopy at baseline, in whom a an endoscopic examination performed during the follow-up for recurrent haemoptysis may allow an aetiological diagnosis | One year
  To evaluate the proportion of patients with a negative bronchoscopy at baseline, in whom a subsequent endoscopic examination performed during the follow-up for recurrent haemoptysis may allow an aetiological (endoscopic and/or microbiological and/or anatomopathological) diagnosis
To evaluate the proportion of patients with a negative chest CT scan and bronchoscopy in whom lung cancer may be diagnosed during the follow-up | One year
  To evaluate the proportion of patients with a negative chest CT scan and bronchoscopy in whom lung cancer may be diagnosed during the follow-up
To evaluate the main clinical characteristics (e.g., severity of haemoptysis) of these patients, the rate and severity of symptom recurrence and the mortality rate after one year of follow-up. | One year
  To evaluate the main clinical characteristics (e.g., severity, duration of haemoptysis) of patients with haemoptysis with negative chest CT scan and bronchoscopy, the rate and severity of symptom recurrence and the mortality rate after one year of follow-up in this cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mondoni, MD, Principal Investigator — Respiratory Unit, ASST Santi Paolo e Carlo, San Paolo Hospital, Milan
Locations (14):
- Italy (13):
  - - Respiratory Unit, ASST Papa Giovanni XVIII, Bergamo
  - - Interventional Pulmonology Unit, Policlinico S. Orsola-Malpighi, Bologna
  - Department of Pulmonary and Critical Care Medicine, Sant'Anna Hospital, Como
  - Respiratory Unit, ASST Lodi, Lodi
  - Respiratory Unit, ASST Santi Paolo e Carlo, Milan
  - - Respiratory Unit, Sacco Hospital, ASST Fatebenefratelli-Sacco, Milan
  - Respiratory Unit, San Gerardo Hospital, ASST Monza, Monza
  - Interventional Pulmonology Unit, Dept of Pulmonology, Oncology and Hematology, Cardarelli Hospital, Naples
  - - Respiratory Unit, IRCCS Foundation Policlinico San Matteo, Pavia
  - Pulmonology Unit, Azienda Unità Sanitaria Locale - IRCCS di Reggio Emilia, Reggio Emilia
  - - Interventional Pulmonology Unit, Policlinico Agostino Gemelli, Roma
  - - Respiratory Unit, A.O.U. Città della Salute e della Scienza di Torino, Torino
  - Department of Pulmonology, University Hospital of Udine (ASUFC), Udine
- Interventional Pulmonology Unit, Respiratory Department, University Hospital Santa Creu i Sant Pau, Barcelona, Spain